CLINICAL TRIAL: NCT05413577
Title: Reducing Parental Stress Via Instant Messaging During COVID-19 Pandemic: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lam Lun Wai Doris, Principal Investigator, Graduate Student in Clinical Psychology, Department of Psychology, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBRE-20-562
Record Dates: First submitted 2022-06-04; First posted 2022-06-10 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Parents; Parenting; Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group was invited to listen to a 15-minute mindfulness instructional recording delivered daily through an instant messaging application and to practice accordingly for 14 consecutive days at their own choice of time and place.
  Interventions: Behavioral: Mindfulness training
- Waitlist control group (No Intervention): The waitlist control group was only be required to complete the demographic information, pre, post experiment and follow-up questionnaires before they receive the mindfulness training intervention.

INTERVENTIONS:
Behavioral: Mindfulness training — The intervention recordings taught the basic concepts of mindfulness through simple guided meditations with content supported by science. Each recording had the same format that included (1) a daily theme, (2) a meditation exercise echoing the theme, (3) a suggested exercise for practice, and (4) an invitation for participants to give a short response to their meditation experience at the end of the recording.
  Arms: Experimental Group

SUMMARY:
This research investigated the effects of mindfulness practice on mental wellbeing and parenting behaviour, with the instruction recordings delivered via existing instant messaging applications, including Whatsapp and Signal. The two-week mindfulness program targeted parents with children in Nursery, Kindergarten to Primary School. Due to the suspension of schools, work from home policies, parents spend increased amount of time with their children. News reports have indicated that with the mounting care taking responsibilities and downturn of economy amidst the epidemic, parents have been experiencing higher stress that may negatively impact their wellbeing and parent-child relationship. This study delivered an app-based intervention that aims at enhancing mindful parenting at the time of corona, where social distancing is emphasized.

ELIGIBILITY:
Inclusion Criteria:

Parents with at least one child who is in Primary School or below.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Parental Stress Scale | Change from Baseline Parental Stress Scale at immediately after the intervention and two weeks after intervention
  The Parental Stress Scale was used to measure self-perceived stress specific to the parenting role. Parental Stress Scale was originally developed by Berry and Jones (1995) to measure parental feelings and experiences in terms of rewards, satisfaction, controllability, and stress. The minimum score was 0 and the maximum score was 64. A score of 0 represents lowest level of parental stress possible, whereas a score of 64 represents highest level of parental stress. Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Well-being WHO 5-item index | Change from Baseline Well-being WHO 5-item index at immediately after the intervention and two weeks after intervention
  Global mental well-being was measured using the Well-being WHO 5-item index (Topp et al., 2015).The minimum score was 0 and the maximum score was 25. A score of 0 represents worst possible, whereas a score of 25 represents best possible quality of life. Higher scores indicate better outcome.
Mindfulness in Parenting Scale | Change from Baseline Interpersonal Mindfulness in Parenting scale at immediately after the intervention and two weeks after intervention
  The 31-item Interpersonal Mindfulness in Parenting scale was adopted to measure parents' self-reported engagement in mindful parenting (Duncan, 2007). The minimum score was 0 and the maximum score was 155. A score of 0 represents lowest level of parental mindfulness, whereas a score of 155 represents highest level of parental mindfulness possible. Higher scores indicate better outcome.
Parent Behavior Inventory | Change from Baseline Parent Behavior Inventory at immediately after the intervention and two weeks after intervention
  The Parent Behavior Inventory was used to assess the change in parenting behavior before and after the intervention. The Parent Behavior Inventory has two independent scales, supportive/engaged and hostile/coercive parenting (Lovejoy et al., 1999), The minimum score was 0 and the maximum score for each scale was 50. A score of 0 represents lowest frequency of parenting behaviors on supportive/engaged and hostile/coercive parenting, whereas a score of 50 represents highest frequency of supportive/engaged and hostile/coercive parenting possible. Higher scores of supportive/engaged scale indicate better outcome. Lower scores of hostile/coercive scale indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lun Wai Doris Lam, M.S.Sc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No identifiable personal information was collected. Surveys were be anonymized to protect the privacy of research participants. All information obtained in the course of this experiment will be used for research purposes only; it will be protected and kept confidential by the researchers of this project and not be shared with a third party unless forced by law.